CLINICAL TRIAL: NCT01239979
Title: Evaluation of the Association Between Myeloperoxidase Levels and Cardiovascular Risk Factors in Patients With Coronary Artery Disease
Brief Title: Plasma Myeloperoxidase Levels in Patients With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Gholam Basati, School of pharmacy and pharmaceutical sciences
Other Study IDs: 388417
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stable, Unstable , control

SUMMARY:
The investigators sought to assess whether plasma myeloperoxidase (MPO) levels differ among patients with stable and unstable CAD patients and control subjects, and correlate with inflammatory and clinical risk factors such as ox-LDL, NO,leptin, adiponectin, sPLA2, Lp-PLA2, homocysteine and 3-nitrotyrosine in the patients.

DETAILED DESCRIPTION:
Elevation of the leukocyte enzyme myeloperoxidase (MPO) in stable coronary artery disease (CAD) patients in contrast to unstable CAD patients is controversial and its relationship with some inflammatory and noninflammatory markers such as oxidized LDL (ox-LDL) and nitric oxide (NO) in the CAD patients has not been evaluated yet. Evaluation of these relationships is the aim of the study.Also the relationships between MPO and some other inflammatory biomarker such as leptin, adiponectin, sPLA2, Lp-PLA2, homocysteine and 3-nitrotyrosine are examined. This study includes 50 stable CAD, 50 unstable CAD patients and 50 controls. Plasma MPO, ox-LDL, leptin, adiponectin, sPLA2 levels are determined using enzyme immunoassay.Homocysteine and 3-nitrotyrosine are measured using HPLC-fluorescence method. Plasma total NO and other risk factors such as lipid profile, hypertension, smoking, diabetes mellitus and familial history of CAD are also determined in the patients. Results are statistically analysed and the association between all markers are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Stable and unstable patients with angiographically documented coronary artery disease.
* Control subjects without angiographically documented coronary artery disease.

All subjects Exclusion Criteria:

* Patients with recent (with in 6 month) myocardial infarction or cardiovascular events,
* surgery (with in 3 month),
* cancer and
* infective or inflammatory diseases were not included in the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects are diagnosed angiographically following chest pain, clinical manifestations or suspected changes on ECG at Isfahan Cardiovascular Research Center in Iran
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Plasma myeloperoxidase levels | 3 month

SECONDARY OUTCOMES:
Clinical risk factors | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Saedzaaldin Samsamshariat, PhD, Study Director — - Clinical Biochemistry Department, School of Pharmacy, Isfahan University of Medical Sciences, Isfahan, Iran
Locations (1):
- Isfahan Cardiovascular Research Center, Isfahan, Isfahan, Iran